CLINICAL TRIAL: NCT03912844
Title: European SIR-Spheres Surgical Registry
Acronym: ESSURE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Köln (Other)
Collaborators: Sirtex Technology Pty LTD, Australia (Unknown)
Responsible Party: Sponsor
Other Study IDs: 18-337
Record Dates: First submitted 2019-04-03; First posted 2019-04-11 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Hepatectomy
Keywords: SIRT; liver resection; hypertrophy; liver metastases; liver transplantation
MeSH Terms: conditions — Hypertrophy | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver resection/liver transplantation after SIRT: The cohort consist of patients that, after decision of a multidisciplinary tumor board have received a SIRT/TARE or will receive a SIRT/TARE to make them later eligible for following liver resection or liver transplantation.
  Interventions: Procedure: SIRT followed by liver resection or liver transplantation

INTERVENTIONS:
Procedure: SIRT followed by liver resection or liver transplantation — The ESSURE registry is a prospective observational study. Patients are only asked to be enrolled when they are treated with SIR-Spheres microspheres followed by liver resection/liver transplantation or when SIRT has been performed with the intention to downsize/ downstage the tumor, to induce hypertrophy of the contralateral lobe, making the patient eligible for a future liver resection/transplantation. In no way will participation in the registry influence the way in which the patient is treated according to the treating clinician, or will it influence the quality of the treatment. If a patient is included in the registry, a documented decision of a multidisciplinary tumour board for the treatment algorithm including SIRT must be available. The follow-up periods depend on the treating clinician and local practice and guidelines. Typically, the follow ups are done every three months. So data of a single patient will be included over two years after the treatment.

SUMMARY:
Liver resection is the only curative treatment option for primary and secondary liver tumors. For some primary or secondary malignancies (HCC, NET) liver transplantation is a possible treatment option. Unfortunately, the majority of patients show a high hepatic tumor load or adverse intrahepatic distribution, that resection or transplantation at the time of initial diagnosis is not possible. In that case different treatment approaches are possible. For those patients that are very unlikely to ever become resectable, palliative systemic therapy is the preferred treatment option. For those patients that may become resectable after downsizing of the tumors or increase of volume of the future liver remnant secondary resection after induction therapy may be a possibility. Then, an induction treatment that has the most likelihood of causing physical shrinkage of the tumors is usually preferred. One of the approaches to create contralateral hypertrophy to increase future liver remnant is portal vein embolization. However, tumor growth might be stimulated during the phase of hypertrophy. Selective internal radiation therapy (SIRT) with SIR-Spheres Y-90 resin microspheres is an endovascular interventional radio-oncologic procedure treating primary and secondary liver tumors1-3. It offers radiation therapy with yttrium-90, a high-energy beta-emitting isotope, directly in the vascular system of liver tumors. It treats the tumor locally, saves healthy liver tissue and could lead to hypertrophy of this residual healthy liver tissue due to the embolization effect. Therefore secondary liver resection after SIRT might become possible4,5. SIRT could also be an option as bridging-, downsizing- or downstaging-therapy before liver transplantation.

Liver resection with local tumor treatment and hypertrophy induction after SIRT seems to be a promising therapy option. Previous reports have shown the feasibility, safety and efficacy of this therapeutic strategy.

Aim of the European SIR-Spheres Surgical Registry - ESSURE - is now to further improve the understanding and optimize the process and patient selection of this therapy strategy in its true clinical setting. This registry enables data collection on the real-life clinical application of liver resection/liver transplantation after SIRT.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Primary or secondary liver tumors
* Treatment of liver tumors with SIR-Spheres Y-90 resin microspheres with the intention to make patient eligible for liver resection/liver transplantation
* Decision of a multidisciplinary tumor board on the patient's therapy regime
* Signed informed-consent form

Exclusion Criteria:

* under 18 years
* not able to sign informed consent
* no decision of a multidisciplinary tumorboard

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are only asked to be enrolled when they are treated with SIR-Spheres microspheres followed by liver resection/liver transplantation or when SIRT has been performed with the intention to downsize/ downstage the tumor, to induce hypertrophy of the contralateral lobe, making the patient eligible for a future liver resection/transplantation. In no way will participation in the registry influence the way in which the patient is treated according to the treating clinician, or will it influence the quality of the treatment. If a patient is included in the registry, a documented decision of a multidisciplinary tumour board for the treatment algorithm including SIRT must be available. The follow-up periods depend on the treating clinician and local practice and guidelines. Typically, the follow ups are done every three months. So data of a single patient will be included over two years after the treatment.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-07-25 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects that receive liver resection/liver transplantation after SIRT | 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Bruns, MD, PhD, Study Chair — Department of General, Visceral and Cancer Surgery, University of Cologne
Locations (1):
- University of Cologne, Department of General, Visceral and Cancer Surgery, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No